CLINICAL TRIAL: NCT05544695
Title: Real-world Evidence Observational Study to Evaluate Performance and Safety of Intravesical Sodium Hyaluronate (Cystistat®) in the Treatment of Patients With Interstitial Cystitis (IC) / Bladder Pain Syndrome (BPS)
Brief Title: Real-world Evidence Study on Cystistat
Acronym: IC/BPS
Status: Completed | Type: Observational
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Other Study IDs: CYST-SLZ-7001
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Interstitial Cystitis and Bladder Pain Syndrome
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: intravesical sodium hyaluronate (Cystistat®) — Cystistat will be instilled into the bladder according to the instructions for use and in line with the routine clinical practice.

SUMMARY:
This study will be conducted with the aim of ensuring the continued acceptability of the benefit-risk ratio and confirming the safety and performance of the device throughout its expected lifetime. Cystistat is supplied as a 50 mL solution containing 40 mg of sodium hyaluronate. It is indicated for the temporary replacement of the GAG layer in the bladder.

DETAILED DESCRIPTION:
Real-world evidence observational studies are considered as an expedient tool to reflect the use of a product under real life conditions.

ELIGIBILITY:
Inclusion Criteria:

* First prescription of Cystistat according to instructions for use.
* Female patients of any ethnic origin with clinical diagnosis of interstitial cystitis (IC)/bladder pain syndrome (BPS). If in accordance with routine clinical practice at the site, ESSIC diagnostic criteria will be used.
* Age: 18 years and older.
* At least 6 months duration of bladder pain/discomfort symptom(s), e.g. constant bladder pain/discomfort or bladder pain/discomfort when voiding or as a burning sensation between voids as the bladder fills with urine.
* At least one accompanying intermittent or persistent lower urinary tract symptom, such as urinary frequency, urgency, or nocturia during the previous 6 months.
* Bladder Pain/ Interstitial Cystitis Symptom Score (BPIC-SS) > 18 prior to first treatment.
* Written informed consent.

Exclusion Criteria:

* Known hypersensitivity reactions to sodium hyaluronate.
* Pregnancy / planned pregnancy or breastfeeding during the course of this NIS.
* Known history of any GAG substitution therapy within the last 2 years.
* Known history of fulguration or resection of Hunner's lesions.
* Known diagnosis of recurrent urinary tract infection or overactive bladder.
* Any other conditions or diseases that can cause similar symptoms, using information from medical history, physical examination findings, laboratory studies (e.g., urine bacterial culture), and other previously performed procedures (e.g., urodynamics, cystoscopy, laparoscopy, radiological studies).
* Patients are not able to fulfil study requirements according to physician's opinion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients of any ethnic origin with clinical diagnosis of interstitial cystitis (IC)/bladder pain syndrome (BPS).
Study Population: Approximately 74 female patients with IC/BPS will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient did not receive study treatment due to withdrawal of consent.
Groups:
- Single Arm: Cystistat® 40 mg/50 mL Solution: All participants received treatment per standard of care
Period: Overall Study
Arm/Group | Single Arm: Cystistat® 40 mg/50 mL Solution
Started | 73
Completed | 68
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm: Cystistat® 40 mg/50 mL Solution
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.9 (17.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Caucasian | 67
  Ethnicity: African | 1
  Ethnicity: Hispanic | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Europe | 73
Bladder Pain/ Interstitial Cystitis Symptom Score [Mean (Standard Deviation); unit: score on a scale] — The Bladder Pain/ Interstitial Cystitis Symptom Score (BPIC-SS) is a validated questionnaire for the measurement of IC/BPS symptoms. It contains 8 questions and the total score ranges from 0 to 38, with higher scores indicating a worse situation. Population: Full analysis set
  score on a scale
    number analyzed (Participants) | 71
    (all) | 29.3 (4.58)
Visual Analogue Scale (urinary urgency) [Mean (Standard Deviation); unit: units on a scale] — Patients will be asked to assess their urinary urgency on the VAS using the question "How intense was urinary urgency over the last 3 days?". The VAS will be an unmarked line ranging from 0 to 100 mm, where 0 = "no urgency" and 100 = "worst possible urgency". Population: Full analysis set
  units on a scale
    number analyzed (Participants) | 71
    (all) | 75.2 (21.70)
Visual Analogue Scale (bladder pain) [Mean (Standard Deviation); unit: units on a scale] — Patients will be asked to assess their bladder pain on the VAS using the question "How was your bladder pain over the last 3 days?". The VAS will be an unmarked line ranging from 0 to 100 mm, where 0 = "no pain" and 100 = "worst possible pain". Population: Full analysis set
  units on a scale
    number analyzed (Participants) | 71
    (all) | 74.7 (18.70)
Visual Analogue Scale (quality of life) [Mean (Standard Deviation); unit: units on a scale] — Patients will be asked to assess QoL on the VAS using the question "How good or bad would you rate your overall health condition throughout the last 3 days?". The VAS will be an unmarked line ranging from 0 to 100 mm, where 0 = "the worst health you can imagine" and 100 = "the best health you can imagine". Population: Full analysis set
  units on a scale
    number analyzed (Participants) | 71
    (all) | 53.1 (28.90)

OUTCOME MEASURES:

1. Primary Outcome: Patient Global Assessment (PGA)
Description: For the primary analysis, a responder was defined as a participant who had an improvement on the PGA scale (i.e., PGA evaluated as markedly improved, moderately improved, or slightly improved. In case of slightly improved, participants were considered as responder only if the question "Did therapy have a positive effect on your life, and would you undergo this treatment again?" is answered with "Yes".).
Time Frame: Up to week 12
Population: Full analysis set
Measure: Number (90% Confidence Interval); unit: percentage of participants (%)
Arm/Group | Single Arm: Cystistat® 40 mg/50 mL Solution
Number analyzed (Participants) | 71
percentage of participants (%) | 90.1 [82.28 to 95.28]

2. Secondary Outcome: Assessment of Bladder Pain/ Interstitial Cystitis Symptom Score
Description: The Bladder Pain/ Interstitial Cystitis Symptom Score (BPIC-SS) is a validated questionnaire for the measurement of IC/BPS symptoms. It contains 8 questions and the total score ranges from 0 to 38, with higher scores indicating a worse situation
Time Frame: Up to week 12 and additionally at Month 6
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale (change from baseline)
Arm/Group | Single Arm: Cystistat® 40 mg/50 mL Solution
Number analyzed (Participants) | 71
score on a scale (change from baseline)
  End of treatment or latest week 12 | -13.8 (8.62)
  Month 6 | -15.3 (9.15)

3. Secondary Outcome: Assessment of Visual Analogue Scale (VAS) for Bladder Pain
Description: Patients will be asked to assess their bladder pain on the VAS using the question "How was your bladder pain over the last 3 days?". The VAS will be an unmarked line ranging from 0 to 100 mm, where 0 = "no pain" and 100 = "worst possible pain".
Time Frame: Up to week 12 and additionally at Month 6
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: units on a scale (change from baseline)
Arm/Group | Single Arm: Cystistat® 40 mg/50 mL Solution
Number analyzed (Participants) | 71
units on a scale (change from baseline)
  End of treatment or latest week 12 | -42.0 (27.49)
  Month 6 | -49.2 (29.69)

4. Secondary Outcome: Assessment of Visual Analogue Scale (VAS) for Urinary Urgency.
Description: Patients will be asked to assess their urinary urgency on the VAS using the question "How intense was urinary urgency over the last 3 days?". The VAS will be an unmarked line ranging from 0 to 100 mm, where 0 = "no urgency" and 100 = "worst possible urgency".
Time Frame: Up to week 12 and additionally at Month 6
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: units on a scale (change from baseline)
Arm/Group | Single Arm: Cystistat® 40 mg/50 mL Solution
Number analyzed (Participants) | 71
units on a scale (change from baseline)
  End of treatment or latest week 12 | -39.3 (28.90)
  Month 6 | -49.2 (30.48)

5. Secondary Outcome: Assessment of Visual Analogue Scale (VAS) for Quality of Life (QoL)
Description: Patients will be asked to assess QoL on the VAS using the question "How good or bad would you rate your overall health condition throughout the last 3 days?". The VAS will be an unmarked line ranging from 0 to 100 mm, where 0 = "the worst health you can imagine" and 100 = "the best health you can imagine".
Time Frame: Up to week 12 and additionally at Month 6
Population: Full anaylsis set
Measure: Mean (Standard Deviation); unit: units on a scale (change from baseline)
Arm/Group | Single Arm: Cystistat® 40 mg/50 mL Solution
Number analyzed (Participants) | 71
units on a scale (change from baseline)
  End of treatment or latest week 12 | 17.1 (35.84)
  Month 6 | 27.2 (33.27)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Single Arm: Cystistat® 40 mg/50 mL Solution: Per standard of care
Arm/Group | Single Arm: Cystistat® 40 mg/50 mL Solution
All-Cause Mortality (participants affected / at risk) | 0/73
Serious Adverse Events (participants affected / at risk) | 1/73
Other Adverse Events (participants affected / at risk) | 13/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm: Cystistat® 40 mg/50 mL Solution (N=73)
pyrexia (General disorders) | 1 (1) — non-related SAE
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm: Cystistat® 40 mg/50 mL Solution (N=73)
Catheter Site Pain (General disorders) | 2 (2)
Abdominal Pain Lower (Gastrointestinal disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Condition Agravated (General disorders) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 3 (3)
Dysuria (Renal and urinary disorders) | 2 (3)
Renal Colic (Renal and urinary disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT05544695/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT05544695/SAP_001.pdf